CLINICAL TRIAL: NCT01282645
Title: A Retrospective Case Series to Evaluate the Long Term Outcome of the Use of Synthes Patient Specific Implants (PSI®) Made of Polyether Ether Ketone (PEEK) for the Treatment of Cranial Defects in Patients With a Mature Skeleton
Brief Title: Case Series to Evaluate Patient Specific Implants (PSI) in Polyether Ether Ketone (PEEK) Performance After 2 Years
Status: Withdrawn | Type: Observational
Sponsor: Synthes GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: STU-CMF-C-16-204-01
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: E04.525.190; Craniotomy; Craniectomy
Keywords: Cranial defect; PSI; patient specific implant; PEEK; polyether ether ketone; craniectomy; craniotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PSI in PEEK: All study subjects have received a Patient Specific Implant (PSI) made of PEEK to repair a cranial defect
  Interventions: Device: PSI in PEEK

INTERVENTIONS:
Device: PSI in PEEK — A Patient Specific Implant made of Polyether Ether Ketone to repair a cranial defect
  Other Names: Patient Specific Implant in Polyether Ether Ketone

SUMMARY:
The primary objective of this retrospective study is to evaluate the percentage of patients with device related adverse events (infection, rejection, dislocation, fracture of the implant) in the first 24 months after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18 years or over at the time of inclusion into the study
* Received a Synthes PSI® made of PEEK intended for replacement of bony voids in the cranial/craniofacial skeleton at least 24 months before inclusion in the study
* Ability to obtain written informed consent from the recipient or the recipient's legal guardian
* Ability to comply with the procedures described in the protocol, including responding to simple questionnaires either by the recipient in person or by a next relative (spouse, parent) who lives with the recipient

Exclusion Criteria:

* Patient was contraindicated to receive a PSI made of PEEK at the time of implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In 30 clinics worldwide, all patients who received a PSI in PEEK at least 2 years ago, who fullfil the in-and exclusion criteria, will be asked to participate
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Device related adverse events | 0-24 months post initial implantation
  Percentage of patients with the following device related adverse events:
  * infection
  * rejection
  * dislocation
  * fracture

SECONDARY OUTCOMES:
Explantation | 0 months - study visit at least 24 months after implantation (or scheduled up to 3 months after the study visit)
  Explantation, as a result of a device-related adverse event or for another reason
Cosmetic result | surgery - at discharge
  Evaluation of the cosmetic result by the surgeon by means of a VAS 0-100, immediately after the surgery or until the patient was discharged from the hospital (any timepoint available)
Cosmetic result | at the study visit, which is at least 24 months after implantation
  Evaluation of the cosmetic result by the surgeon by means of a VAS 0-100, during the study visit, at least 24 months after implantation (see inclusion criteria)
Clinical result | surgery - at discharge
  Evaluation of the clinical result by the surgeon by means of a VAS 0-100, immediately after the surgery or until the patient was discharged from the hospital (any timepoint available)
Clinical result | At the study visit, which is at least 24 months after implantation
  Evaluation of the cosmetic result by the surgeon by means of a VAS 0-100, during the study visit, at least 24 months after implantation (see inclusion criteria)
Pressure sensitivity | At the study visit, which is at least 24 months after implantation
  Evaluation of the pressure sensitivity by the patient (or next of kin appreciation in case of severe disability) by means of a VAS 0-100, during the study visit, at least 24 months after implantation (see inclusion criteria)
Heat / cold sensitivity | At the study visit, which is at least 24 months after implantation
  Evaluation of the heat/cold sensitivity by the patient (or next of kin appreciation in case of severe disability) by means of a VAS 0-100, during the study visit, at least 24 months after implantation (see inclusion criteria)
Cosmetic result | At the study visit, which is at least 24 months after implantation
  Evaluation of the cosmetic result by the patient (or next of kin in case of severe disability) by means of a VAS 0-100, during the study visit, at least 24 months after implantation (see inclusion criteria)
Event-free survival | 0 months - at the study visit, which is at least 24 months after implantation
  Number of months of event-free survival, in terms of device related adverse events:
  * Infection (superficial and/or deep) [Time frame 0 months - study visit]
  * Rejection of the implant [Time frame 0 months - study visit]
  * Dislocation of the implant [Time frame 0 months - study visit]
  * Fracture of the implant [Time frame 0 months - study visit]

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lauwers, MD, Principal Investigator — Centre Hospitalier Universitaire de Toulouse, Toulouse, France
Locations (30):
- AKH Allgemeines Krankenhaus, Vienna, Austria
- Hôpital Erasme ULB, Brussels, Belgium
- Chile (2):
  - Hospital San Pablo de Coquimbo, Coquimbo
  - Hospital de Trabajador de Santiago, Santiago
- Colombia (4):
  - Hospital San José, Bogotá
  - Hospital Universitario San Ignacio, Bogotá
  - Instituto Roosevelt, Bogotá
  - Hospital Universitario del Valle, Santiago de Cali
- Hospital Clinica Biblica, Cartago, Costa Rica
- University Hospital, Ostrava, Czechia
- Rigshospital, Copenhagen, Denmark
- Oulu University Hospital, Oulu, Finland
- Centre Hospitalier Universitaire, Toulouse, France
- Germany (5):
  - Universitätsklinikum Aachen, Aachen
  - HELIOS-Klinikum Emil von Behring, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Clemenshospital Münster, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
- Hospital da Universidade, Coimbra, Portugal
- National Neuroscience Institute, Singapore, Singapore
- Spain (3):
  - Hospital 12 de Octubre, Madrid
  - Ramon y Cajal Hospital, Madrid
  - Clinica Universitaria Navarra, Pamplona
- Switzerland (5):
  - Inselspital, Bern
  - Hôpital Cantonal Universitaire, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital St- Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich
- United Kingdom (2):
  - Queen Victoria Hospital, East Grinstead
  - The Walton Center, Liverpool